CLINICAL TRIAL: NCT01163487
Title: Phase I Trial of Metabolic Reprogramming Therapy for Treatment of Recurrent Head and Neck Cancers
Brief Title: Metabolic Reprogramming Therapy for Treatment of Recurrent Head and Neck Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel T. Chang (Other)
Responsible Party: Sponsor-Investigator, Daniel T. Chang, Assistant Professor of Radiation Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-18245; SU-05052010-5866 (Other: Stanford University); ENT0031 (Other: OnCore)
Record Dates: First submitted 2010-07-06; First posted 2010-07-15 (Estimated); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Head and Neck Cancer; Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dichloroacetate (DCA) (Experimental): 25 mg/kg/day, 37.5 mg/kg, or 50 mg/kg/day oral DCA.
  Interventions: Drug: Dichloroacetate; Device: EF5

INTERVENTIONS:
Drug: Dichloroacetate — 25-50mg/kg per day; oral
  Other Names: DCA
Device: EF5 — 21 mg/kg; IV
  Other Names: EF-5

SUMMARY:
The purpose of this study is to study the effect of the drug DCA (dichloroacetate) on recurrent head and neck cancers. Part of this study will also use EF5 PET scan to study tumor hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed head and neck squamous cell carcinoma
* Age > 18 years old
* Patients must have unresectable disease in which there is no accepted potentially curative treatment option
* Patients must have acceptable organ and marrow function as defined below:
* leukocytes >3,000/uL
* absolute neutrophil count >1,500/uL
* platelets >90,000/uL
* total bilirubin <=1.5X normal institutional limits
* AST(SGOT)/ALT(SGPT) <=2.5 X normal institutional limits with the following exceptions:

  1. Patients with documented tumors involving the liver who have Grade <2 elevations in AST, ALT, and/or alkaline phosphatase are eligible if <5X ULN.
  2. Patients with documented tumors involving bone who have a Grade <2 elevation in alkaline phosphatase are eligible if <5X ULN.
* creatinine <=1.5X normal institutional limits OR creatinine clearance >50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation
* Patients must have non-cranial gross disease that is greater than 1 cm on CT scan prior to enrollment
* Disease must be FDG-avid on PET scanning
* Creatinine within normal institutional limits
* Eastern Clinical Oncology Group performance status 0, 1 or 2 (Appendix 1)
* Life expectancy > 12 weeks
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Women who are pregnant
* Administration of any systemic cytotoxic agents within the last 2 weeks of enrollment
* Patients who are unwilling or unable to provide informed consent
* Patients who have potentially curable disease
* Participation in another concurrent treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-08; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of DCA in patients with recurrent head and neck cancer who have failed first-line therapy. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2015-01-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT01163487/ICF_000.pdf